CLINICAL TRIAL: NCT04097028
Title: Use of Trifluridine/Tipiracil (TAS-102) and Oxaliplatin as Induction Chemotherapy in Resectable Esophageal and Gastroesophageal Junction (GEJ) Adenocarcinoma
Brief Title: Use of Trifluridine/Tipiracil and Oxaliplatin as Induction Chemotherapy for the Treatment of Resectable Esophageal or Gastroesophageal Junction (GEJ) Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Comprehensive Cancer Network (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 443819
Record Dates: First submitted 2019-09-18; First posted 2019-09-20 (Actual); Results first posted 2024-01-18 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-03

CONDITIONS: Clinical Stage IIA Esophageal Adenocarcinoma AJCC v8; Clinical Stage IIA Gastroesophageal Junction Adenocarcinoma AJCC v8; Clinical Stage III Esophageal Adenocarcinoma AJCC v8; Clinical Stage III Gastroesophageal Junction Adenocarcinoma AJCC v8; Clinical Stage IVA Esophageal Adenocarcinoma AJCC v8; Clinical Stage IVA Gastroesophageal Junction Adenocarcinoma AJCC v8; Pathologic Stage IIB Esophageal Adenocarcinoma AJCC v8; Pathologic Stage IIB Gastroesophageal Junction Adenocarcinoma AJCC v8; Pathologic Stage III Esophageal Adenocarcinoma AJCC v8; Pathologic Stage III Gastroesophageal Junction Adenocarcinoma AJCC v8; Pathologic Stage IIIA Esophageal Adenocarcinoma AJCC v8; Pathologic Stage IIIA Gastroesophageal Junction Adenocarcinoma AJCC v8; Pathologic Stage IIIB Esophageal Adenocarcinoma AJCC v8; Pathologic Stage IIIB Gastroesophageal Junction Adenocarcinoma AJCC v8; Pathologic Stage IVA Esophageal Adenocarcinoma AJCC v8; Pathologic Stage IVA Gastroesophageal Junction Adenocarcinoma AJCC v8
MeSH Terms: interventions — Trifluridine; trifluridine tipiracil drug combination; Thymidine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (TAS-102, oxaliplatin) (Experimental): Patients receive oxaliplatin IV over 2 hours on day 1 and trifluridine and tipiracil hydrochloride PO BID on days 1-5. Treatment repeats every 14 days for 3 cycles in the absence of disease progression or unacceptable toxicity. Patients then undergo standard of care chemoradiation therapy followed by surgery.
  Interventions: Drug: Trifluridine and Tipiracil Hydrochloride; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Trifluridine and Tipiracil Hydrochloride — Given PO
  Other Names: 733030-01-8; Lonsurf; TAS 102; Thymidine; Mixt. with 5-Chloro-6-((2-imino-1-pyrrolidinyl)methyl)-2,4(1H,3H)-pyrimidinedione Monohydrochloride; Tipiracil Hydrochloride Mixture with Trifluridine; Trifluridine/Tipiracil
Drug: Oxaliplatin — Given IV
  Other Names: 1-OHP; 266046; 61825-94-3; [(1R,-2R)-1,2-cyclohexanediamine-N,N''][oxalato (2--)-O,O'']platinum; Ai Heng; Aiheng; Dacotin; Dacplat; Diaminocyclohexane Oxalatoplatinum; Eloxatin; Eloxatine; JM-83; oxalato (1R,2R-cyclohexanediamine)platinum(II); oxalato (trans-l-1,2-diaminocyclohexane)platinum(II); Oxalatoplatin; OXALIPLATIN,; RP 54780; RP-54780; SR-96669; trans-l DACH oxalatoplatinum

SUMMARY:
This phase II trial studies how well trifluridine/tipiracil and oxaliplatin work as the first line of treatment (induction) in treating patients with esophageal or gastroesophageal junction adenocarcinoma that can be removed by surgery (resectable). Drugs used in chemotherapy, such as trifluridine/tipiracil and oxaliplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

-Evaluate the pathologic complete response (path CR) rate in participants with esophageal and gastroesophageal junction (GEJ) adenocarcinoma when trifluridine and tipiracil hydrochloride (trifluridine/tipiracil [TAS-102]) and oxaliplatin are used as induction chemotherapy prior to surgical resection.

SECONDARY OBJECTIVES:

* Evaluate the 2-year disease-free survival (DFS) and the 2-year overall survival (OS)
* To determinate the safety and tolerability of induction chemotherapy with trifluridine/tipiracil (TAS 102) and oxaliplatin followed by standard chemoradiation and surgery
* Evaluate the metabolic response to induction chemotherapy with TAS 102 and oxaliplatin in participants with esophageal and gastroesophageal junction (GEJ) adenocarcinoma prior to standard chemoradiation and surgical resection

EXPLORATORY OBJECTIVE:

-Correlate circulating tumor deoxyribonucleic acid (DNA) levels with disease recurrence and metabolic response on positron emission tomography (PET) computed tomography (CT).

OUTLINE:

Patients receive oxaliplatin intravenously (IV) over 2 hours on day 1 and trifluridine and tipiracil hydrochloride orally (PO) twice daily (BID) on days 1-5. Treatment repeats every 14 days for 3 cycles in the absence of disease progression or unacceptable toxicity. Patients then undergo standard of care chemoradiation therapy followed by surgery.

After completion of study treatment, patients are followed up every 3-6 months for years 1-2, every 6-12 months.

ELIGIBILITY:
Inclusion Criteria:

* Must have histologically proven loco-regional esophageal or gastroesophageal junction adenocarcinoma
* Endoscopic ultrasound (EUS), or clinically determined node-positive disease with any T-stage or T3-T4a with any N stage: Patients with EUS T4b and any M1 cancer will not be included
* Must have potentially resectable disease
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Hemoglobin >= 9 g/dL
* Absolute neutrophil count >= 1500/mm^3
* Platelet count >= 100,000/mm^3
* Creatinine < 1.5 upper limit of normal (ULN)
* Bilirubin < 1.5 x ULN
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 3 x ULN
* Capacity to take oral tablet(s) without difficulty
* Participants of child-bearing potential must agree to use highly effective contraceptive methods (e.g., hormonal plus barrier method of birth control; abstinence) prior to study entry. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Participant must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Prior chemotherapy, thoracic radiotherapy or prior surgical resection for an esophageal tumor
* Participants with known metastatic disease
* Any concurrent active malignancy that requires active systemic intervention
* Grade 2 or higher peripheral neuropathy
* Participants who have had major surgery or field radiation within 4 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Received an investigational agent within 4 weeks prior to enrollment
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Grade 3 or higher hypersensitivity reaction to oxaliplatin or grade 1-2 hypersensitivity reaction to oxaliplatin not controlled with premedication
* Patient previously treated by TAS 102 or history of allergic reactions attributed to compounds of similar composition to TAS 102 or any of its excipients
* Hereditary problems of galactose intolerance; e.g., Lapp lactase deficiency or glucose galactose malabsorption
* Pregnant or nursing female participants
* Unwilling or unable to follow protocol requirements
* Any condition which in the investigator's opinion deems the participant an unsuitable candidate to receive study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-12-20 (Actual); Primary Completion 2022-12-16 (Actual); Study Completion 2025-02-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christos Fountilas, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (2):
- United States (2):
  - Roswell Park Cancer Institute, Buffalo, New York
  - Stephenson Oklahoma Cancer Center at the University of Oklahoma Health Science Center, Oklahoma City, Oklahoma

REFERENCES:
- [Derived] Mukherjee S, Fujiwara Y, Fountzilas C, Pattnaik H, Chatley S, Vadehra D, Kukar M, Attwood K, George A, Advani S, Yu H, Catalfamo K, Brown A, Spickard E, Fungtammasan A, George S, Liao CY, Iyer R, Hatoum H. Trifluridine/Tipiracil and Oxaliplatin as Induction Chemotherapy in Resectable Esophageal and Gastroesophageal Junction Adenocarcinoma: A Phase II Study. Cancer Med. 2025 Apr;14(7):e70835. doi: 10.1002/cam4.70835. PMID 40200573

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (TAS-102, Oxaliplatin)
Started | 22
Completed | 15
Not Completed | 7
Not completed — Disease Progression Prior to completion of Chemoradiation | 2
Not completed — Adverse Event prior to Completion of Chemoradiation | 2
Not completed — Disease Progression prior to Surgery | 2
Not completed — Adverse Event prior to Surgery | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (TAS-102, Oxaliplatin)
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.7 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 19
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With a Pathologic Complete Response
Description: Will be determined by pathologic examination of resected specimen: complete response to induction chemotherapy followed by standard chemoradiation and surgery. Will be summarized using frequencies and relative frequencies. Will be estimated using an 80% confidence interval obtained using Jeffrey's prior method.
  Response is assessed by the tumor regression score (as proposed by NCCN guidelines):
  Complete Response: No viable cancer cells, including lymph nodes Near Complete Response: Single cells or rare small groups of cancer cells Partial Response: Residual cancer with evident tumor regression but more than single cells or rare small groups of cancer cells Poor or No Response: Extensive residual disease with no evident tumor regression
Time Frame: Assessed at the time of surgery (approximately 6 months after start of neoadjuvant therapy)
Population: Only 15 patients completed surgery.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (TAS-102, Oxaliplatin)
Number analyzed (Participants) | 15
Participants | 2

2. Secondary Outcome: Median Progression Free Survival
Description: Will be summarized using standard Kaplan-Meier methods; where estimates of median survival and two-year survival rates will be obtained with 95% confidence intervals. Progression is assessed by RECIST v1.0, defined as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Time from treatment until disease progression, death from disease, or last follow-up, assessed up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (TAS-102, Oxaliplatin)
Number analyzed (Participants) | 22
months | 20.3 [5.9 to NA] — Due to the sample size and number of events the upper limit of the confidence interval is not estimable (or NE). This is very common in survival data and should not require additional explanation.

3. Secondary Outcome: Median Overall Survival
Description: Will be summarized using standard Kaplan-Meier methods; where estimates of median survival and two-year survival rates will be obtained with 95% confidence intervals
Time Frame: Time from treatment until death due to any cause or last follow-up, assessed up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (TAS-102, Oxaliplatin)
Number analyzed (Participants) | 22
months | 20.3 [8.6 to NA] — Due to the sample size and number of events, the upper limit of the confidence interval is not estimable.

4. Secondary Outcome: Number of Patients With Grade 3 or Higher Treatment Related Adverse Events
Description: Toxicities and adverse events (as per Common Terminology Criteria for Adverse Events version 5.0) will be summarized by attribution and grade using frequencies and relative frequencies.
Time Frame: Up to 30 days after last dose of study drug, which is a maximum of 210 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (TAS-102, Oxaliplatin)
Number analyzed (Participants) | 22
Participants | 5

ADVERSE EVENTS:
Time Frame: Adverse events were monitored up to 30 days after surgery, which is expected to be 50 days and a maximum of 210 days. All cause mortality was monitored up to two years.
Arm/Group | Treatment (TAS-102, Oxaliplatin)
All-Cause Mortality (participants affected / at risk) | 7/22
Serious Adverse Events (participants affected / at risk) | 3/22
Other Adverse Events (participants affected / at risk) | 17/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (TAS-102, Oxaliplatin) (N=22)
Colonic perforation (Gastrointestinal disorders) | 1 (1)
Anaphylaxis (Immune system disorders) | 1 (1)
Lymph gland infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (TAS-102, Oxaliplatin) (N=22)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Bloating (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 11 (11)
Diarrhea (Gastrointestinal disorders) | 9 (9)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Flatulence (Gastrointestinal disorders) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 13 (13)
Oral dysesthesia (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 8 (8)
Fatigue (General disorders) | 13 (13)
Fever (Gastrointestinal disorders) | 3 (3)
Infusion related reaction (Injury, poisoning and procedural complications) | 4 (4)
Lymphocyte count decreased (Investigations) | 2 (2)
Neutrophil count decreased (Investigations) | 5 (5)
Platelet count decreased (Investigations) | 3 (3)
White blood cell decreased (Investigations) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 6 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Dysesthesia (Nervous system disorders) | 5 (5)
Dysgeusia (Nervous system disorders) | 5 (5)
Headache (Nervous system disorders) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 7 (7)
Insomnia (Psychiatric disorders) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-06): https://cdn.clinicaltrials.gov/large-docs/28/NCT04097028/Prot_SAP_000.pdf